CLINICAL TRIAL: NCT02685111
Title: Intermittent Every Other Days of 5 Shot-filgrastim Compared With Single Pegfilgrastim in Breast Cancer Patients Receiving Adjuvant Docetaxel, Doxorubicin, and Cyclophosphamide Chemotherapy (Intermittent G-CSF 105)
Brief Title: Intermittent G-CSF in Patients With Breast Cancer Receiving Adjuvant Docetaxel, Doxorubicin, and Cyclophosphamide (TAC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Sung-Bae Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AMC 2015-1143
Record Dates: First submitted 2016-02-10; First posted 2016-02-18 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer; Neutropenia; Febrile Neutropenia
Keywords: Breast cancer; Adjuvant; Docetaxel; Adriamycin; Cyclophosphamide; Neutropenia; Filgrastim; Pegfilgrastim
MeSH Terms: conditions — Breast Neoplasms; Neutropenia; Febrile Neutropenia | interventions — Filgrastim; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A. Pegfilgrastim (Active Comparator): D2 once a cycle pegfilgrastim arm
  Interventions: Drug: Peg-filgrastim
- B. Filgrastim (Experimental): Intermittent Every Other Days of 5 Shot (D3-11) filgrastim arm
  Interventions: Drug: Filgrastim

INTERVENTIONS:
Drug: Filgrastim — Filgrastim (Gracinᵀᴹ) is administered at the D3, D5, D7, D9, and D11 of each cycle. A dose of 5 μg/kg/day filgrastim is administered S.C. either as a bolus injection or as a continuous injection. Administer into the outer upper arm, abdomen (except within 2 inches of navel), front middle thigh, or the upper outer buttocks area.
  Other Names: Grasinᵀᴹ pfs inj.
  Arms: B. Filgrastim
Drug: Peg-filgrastim — Pegfilgrastim (Neulastaᵀᴹ) is administered at the D2 of each cycle. A dose of 6mg once a cycle is administered S.C., 24 (± 2) hours after completion of chemotherapy.
  Other Names: Neulastaᵀᴹ pfs inj. 6mg/0.6ml
  Arms: A. Pegfilgrastim

SUMMARY:
To compare the efficacy and safety of Day 2 (D2) once a cycle pegfilgrastim with Intermittent Every Other Days of 5 Shot (D3-11) filgrastim in early breast cancer patients treated with adjuvant Docetaxel, Doxorubicin, and Cyclophosphamide (TAC) regimen

DETAILED DESCRIPTION:
According to manufacturers' recommendations (Amgen: Neupogenᵀᴹ), filgrastim are to start 24 hrs after the last dose of chemotherapy and continue until absolute neutrophil count (ANC) has recovered to within the normal range (or for 14 days). However, for economic and practical reasons and/or patient's convenience, it has been common practice to initiate filgrastim at a later days of cycle and/or administer a shorter course of treatment. Data from several clinical studies have shown that 10-11 days' filgrastim treatment is required for optimal prophylaxis for febrile neutropenia (FN), and data from other cancers shows that suboptimal use of G-CSFs could deteriorate clinical outcomes. However, in two recent randomized study with breast cancer patients undergoing TAC chemotherapy, acceptable incidence (7-18%) of FN was shown with the consecutive 6 or 7-daily filgrastim schemes. Also, although there is theoretical concern that there can be wide fluctuations in the patient's ANC over time in alternate or intermittent filgrastim administration, because there was no difference in clinical outcomes between daily- or intermittent-dose filgrastim schedules in previous literatures, the intermittent every other day of 5 shot-filgrastim scheme would have clinical outcomes comparable with previous consecutive 6 or 7-daily filgrastim schemes in coverage of ANC nadir. Therefore, it can be justified to investigate the non-inferiority of intermittent every other days of 5 shot-filgrastim scheme compared with control arm using of pegfilgrastim on D2.

ELIGIBILITY:
Inclusion Criteria:

* The patients who underwent surgery for pathologically diagnosed early breast cancer (high risk stage II or stage III) or completely resected stage IV, and anticipated to undergo adjuvant chemotherapy with TAC regimen (docetaxel, doxorubicin, and cyclophosphamide)
* The patients satisfying laboratory findings below before the enrollment of clinical trials: A. Absolute Neutrophil Count(ANC) ≥ 1,500/mm³; B. Platelet Count ≥ 100,000/mm³; C. Adequate renal functions (Cr < 1.5 X ULN); and D. Adequate liver function (Bilirubin < 1.5 X ULN, AST/ALT < 2.5 X ULN)
* ECOG Performance status: 0-1
* Cardiac ejection fraction ≥ 50% as measured by MUGA or 2D echocardiography without clinically significant abnormalities
* Voluntarily participated in this study, and written informed consent of the patient

Exclusion Criteria:

* Past history of immunotherapy or chemotherapy
* Past history of autologous stem cell transplantation or bone marrow transplantation
* The patient undergone radiation therapy within 4 weeks after written informed consent
* Patient with any other concurrent malignancies or who are currently cured with past history within 5 years (excluding completely resected stage I early skin cancer)
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Other serious illness or medical conditions inadequate to chemotherapy: A. Unstable cardiac disease (i.e. congestive heart failure, arrhythmia, symptomatic coronary artery disease) despite treatment, myocardial infarction within 6 months prior to study entry; B. History of significant neurological or psychiatric disorders including dementia or seizures; Active uncontrolled infection (viral, bacterial or fungal infection); and D. Other serious medical illnesses
* Known hypersensitivity to any of the study drugs or its ingredients
* Concomitant administration of any other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy.
* Past history of usage of granulocyte-colony stimulating factors
* Patients with a known history of HIV (+) or HCV (+). However, HBV(+) patients who undergo primary prophylaxis are eligible.
* Other serious illness or medical conditions determined by investigator

Ages: 19 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of febrile neutropenia | through the completion of cycle 1-3 (each cycle is 21 days), an average of 9 weeks
  Measured at the completion of cycle 3

SECONDARY OUTCOMES:
Incidence of febrile neutropenia at each cycle | At each cycle 1, 2, and 3 (each cycle is 21 days)
  Measured at the completion of each cycle 1, 2, and 3
Rates of anti-microbial use | through the completion of cycle 1-3 (each cycle is 21 days), an average of 9 weeks
  Measured at the completion of cycle 3
Duration of anti-microbial use | through the completion of cycle 1-3 (each cycle is 21 days), an average of 9 weeks
  Measured at the completion of cycle 3
Cumulative dose of chemotherapeutic agents | through the completion of cycle 1-3 (each cycle is 21 days), an average of 9 weeks
  Measured at the completion of cycle 3
Delay rate of next chemotherapy cycle due to inadequate neutrophil recovery | At each cycle 1, 2, and 3 (each cycle is 21 days)
  Measured at the completion of each cycle 1, 2, and 3
Duration of delay of next chemotherapy cycle due to inadequate neutrophil recovery | At each cycle 1, 2, and 3 (each cycle is 21 days)
  Measured at the completion of each cycle 1, 2, and 3

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Bae Kim, Ph.D., Principal Investigator — Department of Oncology, Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scott SD, Chrischilles EA, Link BK, Delgado DJ, Fridman M, Stolshek BS. Days of prophylactic filgrastim use to reduce febrile neutropenia in patients with non-Hodgkin's lymphoma treated with chemotherapy. J Manag Care Pharm. 2003 Mar-Apr;9(2 Suppl):15-21. doi: 10.18553/jmcp.2003.9.s2.15. PMID 14613340
- [Background] von Minckwitz G, Raab G, Caputo A, Schutte M, Hilfrich J, Blohmer JU, Gerber B, Costa SD, Merkle E, Eidtmann H, Lampe D, Jackisch C, du Bois A, Kaufmann M. Doxorubicin with cyclophosphamide followed by docetaxel every 21 days compared with doxorubicin and docetaxel every 14 days as preoperative treatment in operable breast cancer: the GEPARDUO study of the German Breast Group. J Clin Oncol. 2005 Apr 20;23(12):2676-85. doi: 10.1200/JCO.2005.05.078. PMID 15837982
- [Background] Weycker D, Hackett J, Edelsberg JS, Oster G, Glass AG. Are shorter courses of filgrastim prophylaxis associated with increased risk of hospitalization? Ann Pharmacother. 2006 Mar;40(3):402-7. doi: 10.1345/aph.1G516. Epub 2006 Feb 21. PMID 16492793
- [Background] Holmes FA, Jones SE, O'Shaughnessy J, Vukelja S, George T, Savin M, Richards D, Glaspy J, Meza L, Cohen G, Dhami M, Budman DR, Hackett J, Brassard M, Yang BB, Liang BC. Comparable efficacy and safety profiles of once-per-cycle pegfilgrastim and daily injection filgrastim in chemotherapy-induced neutropenia: a multicenter dose-finding study in women with breast cancer. Ann Oncol. 2002 Jun;13(6):903-9. doi: 10.1093/annonc/mdf130. PMID 12123336
- [Background] Green MD, Koelbl H, Baselga J, Galid A, Guillem V, Gascon P, Siena S, Lalisang RI, Samonigg H, Clemens MR, Zani V, Liang BC, Renwick J, Piccart MJ; International Pegfilgrastim 749 Study Group. A randomized double-blind multicenter phase III study of fixed-dose single-administration pegfilgrastim versus daily filgrastim in patients receiving myelosuppressive chemotherapy. Ann Oncol. 2003 Jan;14(1):29-35. doi: 10.1093/annonc/mdg019. PMID 12488289
- [Background] Koumakis G, Vassilomanolakis M, Barbounis V, Hatzichristou E, Demiri S, Plataniotis G, Pamouktsoglou F, Efremidis AP. Optimal timing (Preemptive versus supportive) of granulocyte colony-stimulating factor administration following high-dose cyclophosphamide. Oncology. 1999;56(1):28-35. doi: 10.1159/000011926. PMID 9885374
- [Background] Martin M, Lluch A, Segui MA, Ruiz A, Ramos M, Adrover E, Rodriguez-Lescure A, Grosse R, Calvo L, Fernandez-Chacon C, Roset M, Anton A, Isla D, del Prado PM, Iglesias L, Zaluski J, Arcusa A, Lopez-Vega JM, Munoz M, Mel JR. Toxicity and health-related quality of life in breast cancer patients receiving adjuvant docetaxel, doxorubicin, cyclophosphamide (TAC) or 5-fluorouracil, doxorubicin and cyclophosphamide (FAC): impact of adding primary prophylactic granulocyte-colony stimulating factor to the TAC regimen. Ann Oncol. 2006 Aug;17(8):1205-12. doi: 10.1093/annonc/mdl135. Epub 2006 Jun 9. PMID 16766587
- [Background] von Minckwitz G, Kummel S, du Bois A, Eiermann W, Eidtmann H, Gerber B, Hilfrich J, Huober J, Costa SD, Jackisch C, Grasshoff ST, Vescia S, Skacel T, Loibl S, Mehta KM, Kaufmann M; German Breast Group. Pegfilgrastim +/- ciprofloxacin for primary prophylaxis with TAC (docetaxel/doxorubicin/cyclophosphamide) chemotherapy for breast cancer. Results from the GEPARTRIO study. Ann Oncol. 2008 Feb;19(2):292-8. doi: 10.1093/annonc/mdm438. Epub 2007 Sep 9. PMID 17846019
- [Background] Papaldo P, Lopez M, Marolla P, Cortesi E, Antimi M, Terzoli E, Vici P, Barone C, Ferretti G, Di Cosimo S, Carlini P, Nistico C, Conti F, Di Lauro L, Botti C, Di Filippo F, Fabi A, Giannarelli D, Calabresi F. Impact of five prophylactic filgrastim schedules on hematologic toxicity in early breast cancer patients treated with epirubicin and cyclophosphamide. J Clin Oncol. 2005 Oct 1;23(28):6908-18. doi: 10.1200/JCO.2005.03.099. Epub 2005 Aug 29. PMID 16129844